CLINICAL TRIAL: NCT01275755
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2 Study to Evaluate the Efficacy and Safety of ADL5945 Once Daily for the Treatment of Opioid-induced Constipation in Adults Taking Opioid Therapy for Chronic Noncancer Pain
Brief Title: Evaluation of the Efficacy and Safety of ADL5945 Once Daily for the Treatment of Opioid-induced Constipation in Adults Taking Opioid Therapy for Chronic Noncancer Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2402-002; 45CL243 (Other: Cubist Study Number)
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-10

CONDITIONS: Constipation
Keywords: opioid therapy; constipation; chronic noncancer pain; mu opioid receptor antagonist; ADL5945; Opioid Induced Constipation
MeSH Terms: conditions — Constipation; Opioid-Induced Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Each participant received 1 placebo capsule orally every day (QD) during the Run-in Placebo Period (1 week), the Double-blind Treatment Period (4 weeks), and the Run-out Placebo Period (1 week).
  Interventions: Drug: Placebo
- ADL5945 0.25 mg (Experimental): During the Run-in Placebo Period, each participant received 1 placebo capsule orally QD for 1 week. Then during the Double-blind Treatment Period, each participant received one 0.25-milligrams (mg) ADL5945 capsule orally QD for 4 weeks. Then during the Run-out Placebo Period, each participant received 1 placebo capsule orally QD for 1 week.
  Interventions: Drug: Placebo; Drug: ADL5945 0.25 mg

INTERVENTIONS:
Drug: Placebo
Drug: ADL5945 0.25 mg
  Arms: ADL5945 0.25 mg

SUMMARY:
Morphine and related opioid analgesics are known to slow gastrointestinal (GI) motility and reduce intestinal secretion through their binding to μ opioid receptors (MORs) within the GI tract. The most common symptoms associated with the effects of opioids are constipation and nausea and/or vomiting. Moreover, constipation is a common and distressing side effect of long-term opioid therapy.

The primary objective of this study was to compare ADL5945 once daily, a MOR antagonist, with placebo in the treatment of opioid-induced constipation (OIC) in adults taking long-term opioid therapy for chronic noncancer pain.

ELIGIBILITY:
Key Inclusion Criteria

* be a man or woman aged 18 to 75 years, inclusive, at the time of screening
* have a body weight ≥45 kilograms (kg) and a body mass index (BMI) ≤40 kilograms per square meter (kg/m^2)
* be taking a stable daily dose of opioids of ≥30-milligrams (mg) morphine-equivalent total -daily dose for chronic noncancer pain for ≥30 days before screening
* have opioid-induced constipation (OIC) by history. Additionally, based on the data collected during the 1-week screening period, participants must have <3 spontaneous bowel movements (SBMs) per week and have experienced ≥1 other bowel movement (BM) symptom (that is, straining to pass a stool, lumpy hard stools or small pellets, or sense of incomplete evacuation after passing a stool) for ≥25% of the total BMs
* be willing to discontinue use of all laxatives and stool softeners during the study period except as allowed by the protocol

Key Exclusion Criteria

* be pregnant, lactating, or planning to become pregnant during the study
* have aspartate aminotransferase (AST), alanine aminotransferase (ALT), blood urea nitrogen, or serum creatinine results ≥2 times the upper limit of normal
* have a recent history of myocardial infarction (MI) or unstable angina
* have an active malignancy of any type
* be taking opioids primarily for fibromyalgia
* be taking methadone as a maintenance medication (participants taking methadone for pain may be enrolled)
* be taking intrathecal opioids for the management of pain
* be taking tramadol, tapentadol, or any mixed agonist/antagonist opioid analgesics as the sole opioid for analgesia
* be taking any μ-opioid receptors (MOR) antagonist, including opioids in combination with naloxone, naltrexone, or methylnaltrexone bromide
* be taking medical marijuana
* have gastrointestinal (GI) or pelvic disorders known to affect bowel transit, produce GI obstruction, or contribute to bowel dysfunction
* have taken antispasmodics, antidiarrheals, or prokinetics within 7 days before the start of the screening week
* be taking nonopioid medications known to cause constipation
* be taking antidiarrheals and have an incidence or a history of intermittent diarrhea or loose stools
* be unwilling to abstain from grapefruit and grapefruit-containing products
* have a history of alcoholism or illicit drug dependence or abuse within 5 years before screening
* have positive results on a urine drug screen (excluding opioids) that indicate illicit drug use

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2011-01-19 (Actual); Primary Completion 2011-07-15 (Actual); Study Completion 2011-07-15 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Period: Run-in Placebo Period
Arm/Group | Placebo | ADL5945 0.25 mg
Started | 41 | 40
Completed | 41 | 40
Not Completed | 0 | 0
Period: Double-blind Treatment Period
Arm/Group | Placebo | ADL5945 0.25 mg
Started | 41 | 40
Received at Least 1 Dose of Study Drug | 41 | 40
Completed | 39 | 37
Not Completed | 2 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Period: Run-out Placebo Period
Arm/Group | Placebo | ADL5945 0.25 mg
Started | 39 | 37
Completed | 38 | 37
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug
Groups:
- Placebo: Each participant received 1 placebo capsule orally QD during the Run-in Placebo Period (1 week), the Double-blind Treatment Period (4 weeks), and the Run-out Placebo Period (1 week).
- ADL5945 0.25mg: During the Run-in Placebo Period, each participant received 1 placebo capsule orally QD for 1 week. Then during the Double-blind Treatment Period, each participant received one 0.25-mg ADL5945 capsule orally QD for 4 weeks. Then during the Run-out Placebo Period, each participant received 1 placebo capsule orally QD for 1 week.
- Total: Total of all reporting groups
Arm/Group | Placebo | ADL5945 0.25mg | Total
Number analyzed (Participants) | 41 | 40 | 81
Age, Categorical [Count of Participants; unit: Participants]
  LTE18 | 0 | 0 | 0
  BTWN | 37 | 35 | 72
  GTE65 | 4 | 5 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 56
  Male | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Weekly Average of Spontaneous Bowel Movements (SBMs) During Treatment
Description: An SBM was defined as a bowel movement (BM) with no laxative use in the previous 24 hours. Each weekly SBM average was calculated as follows: (7 × number of SBMs) / (number of days with nonmissing data). The overall SBM rate for the 4-week double-blind treatment period was calculated as follows: (the average of the first week + the average of the second week + the average of the third week + the average of the fourth week) / 4.
Time Frame: Baseline, Weeks 1 through 4 of treatment
Population: All participants who were randomized to study treatment and had at least 1 evaluable SBM post-dose measurement during the Double-blind Treatment Period. Last-observation-carried-forward (LOCF) was used to impute missing postbaseline values.
Measure: Mean (Standard Error); unit: Number of SBMs/week
Groups:
- ADL5945 0.25 mg: During the Run-in Placebo Period, each participant received 1 placebo capsule orally QD for 1 week. Then during the Double-blind Treatment Period, each participant received one 0.25-mg ADL5945 capsule orally QD for 4 weeks. Then during the Run-out Placebo Period, each participant received 1 placebo capsule orally QD for 1 week.
Arm/Group | Placebo | ADL5945 0.25 mg
Number analyzed (Participants) | 41 | 40
Number of SBMs/week | 1.40 (0.26) | 2.58 (0.34)

ADVERSE EVENTS:
Arm/Group | Placebo | ADL5945 0.25 mg
Serious Adverse Events (participants affected / at risk) | 0/41 | 1/40
Other Adverse Events (participants affected / at risk) | 11/41 | 10/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=41) | ADL5945 0.25 mg (N=40)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1) — This Serious Adverse Event occurred 35 days following last dose of double-blind study medication. The participant died as a result of this SAE
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=41) | ADL5945 0.25 mg (N=40)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 3 (3) | 2 (2)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other